CLINICAL TRIAL: NCT05306470
Title: Ethyl Chloride-Endo Ice Versus 5% Lidocaine for Topical Anesthesia of Oral Mucosa - a Randomized Clinical Trial
Brief Title: Ethyl Chloride Versus 5% Lidocaine for Topical Anesthesia of Oral Mucosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Hira Abbasi, Principal Investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Local Anesthetic
Record Dates: First submitted 2022-03-15; First posted 2022-04-01 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Pain; Symptomatic Irreversible Pulpitis
MeSH Terms: conditions — Pain | interventions — Ethyl Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ethyl chloride (Experimental): Pre cooling done by the application of single spray ethyl chloride on a cotton pellet and placed for 30 seconds at the injection site for numbing effect
  Interventions: Procedure: Ethyl chloride
- 5% lidocaine gel (Experimental): 5% lidocaine gel 2ml applied on a cotton pallet for 30 seconds on the oral mucosa at the site of injection for the numbing effect
  Interventions: Procedure: 5% lidocaine gel
- control (No Intervention): Local anesthesia infiltration is administrated without using any numbing agent

INTERVENTIONS:
Procedure: Ethyl chloride — Application of ethyl chloride for a cooling effect to numb the area for oral infiltration anesthetic
  Arms: Ethyl chloride
Procedure: 5% lidocaine gel — Application of 5% lidocaine gel to numb the area for oral infiltration anesthetic
  Arms: 5% lidocaine gel

SUMMARY:
Local anesthesia in the oral cavity is a pain full experience for the patient. All means should be made to reduce the pain and anxiety of the patient for needle stick procedures. My study aims in elevating the pain experienced by the patient during this procedure by using either cold application with ethyl chloride or 5% lidocaine gel.

DETAILED DESCRIPTION:
Local anesthetic procedure is always a dreadful experience for the patient specially for the patients who are already in pain . It is a job of the dentist to provide a painless dental treatment from the very beginning. Most dental procedures require administration of local anesthesia for a painless procedure with local anesthesia procedure being painful itself with the administration of needle in the oral cavity. Dentist everyday in their practice utilise various techniques and procedures in alleviating this painful experience with either application of lidocaine gel or spray . Numbing the oral mucosa with cold application is well documented and tested therefore my study aims in application of ethyl chloride spray on cotton pallet for a duration of 30 seconds in producing the desired numbing effect of the oral mucosa before infiltration of local anesthesia in alleviating the needle prick sensation perceived by the patient.

Pain level is assigned to one of four categorical scores using visual analogue scale

1. :None(0)
2. : Mild (1-3)
3. : Moderate (4-6)
4. : Severe (7-10)

ELIGIBILITY:
Inclusion Criteria:

* No medical history
* No age restrictions
* Patients suffering from Symptomatic Irreversible Pulpitis requiring buccal infiltration

Exclusion Criteria:

* Patients having any medical conditions considered to affect patient safety or the quality of the study
* if they had any known hypersensitivity to local anaesthetics of amide type or any of the other contents in the substance used

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Post oral local anesthetic infiltration pain | immediately after completion of administration of oral local anesthetic infiltration within 60 seconds
  Post administration of oral local anesthetic infiltration pain will be measured by using Visual Analogue Scale(VAS) which is an 10-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured

CONTACTS AND LOCATIONS:
Locations (1):
- Hira Danish, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No